CLINICAL TRIAL: NCT07155031
Title: Kinetics of Pathogen Reduced Red Blood Cell Clearance in Subjects Undergoing Red Cell Exchange for Sickle Cell Disease
Brief Title: Biotin-Acridine Red Cell Exchange Kinetics
Acronym: BARK
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLI 00185
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: pathogen reduction; sickle cell disease; red cell exchange; biotin
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Prospective, Phase 2, non-randomized, open-label, single arm, single center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention Arm (Experimental): All subjects enrolled in CLI00185 will participate in the intervention arm which includes transfusion of a single pathogen reduced red blood cell unit in conjunction with two sequential red cell exchange episodes (as prescribed by subjects attending physician). Subjects will also receive aliquots of biotin labeled red blood cells during the first of the two red cell exchange episodes.
  Interventions: Device: Pathogen reduced red blood cells

INTERVENTIONS:
Device: Pathogen reduced red blood cells — pathogen reduced red blood cells with biotin labeled aliquots will be transfused as part of routine care red cell exchange procedures
  Other Names: Biotin

SUMMARY:
The primary objective of the study is to describe the recovery and survival of pathogen-reduced (PR) red blood cells (RBCs) prepared and stored with the INTERCEPT Blood System for RBCs® (hereafter referred to as INTERCEPT RBCs) in patients with sickle cell disease (SCD) undergoing red cell exchange (RCE) therapy, utilizing flow cytometry for biotin and acridine RBC surface markers.

DETAILED DESCRIPTION:
This trial is designed as a prospective, Phase 2, non-randomized, open-label, single arm, single center study in at least five (5) patients with sickle cell disease (SCD) undergoing red cell exchange (RCE) therapy.

Subjects receiving routine care for SCD utilizing regular RCE therapy at Grady Memorial Healthcare will be approached by Emory investigators and asked to enroll in the trial. Interested subjects will complete an informed consent form (ICF) and undergo pre-study screening, including a test for the presence of naturally-occurring antibodies with specificity for INTERCEPT RBCs and for antibodies with specificity for biotin. Subjects with a positive screen for INTERCEPT RBC antibodies or for biotin antibodies will be excluded from the study. Investigators will screen the current pool of patients receiving RCE treatment at Grady Memorial Healthcare to identify at least five (5) subjects who meet the study's enrollment criteria.

Enrolled and consented subjects will receive a full unit of INTERCEPT RBCs following each of two sequential RCE episodes (RCE #1 and RCE #2). The INTERCEPT RBCs will be administered by simple transfusion immediately following the end of each RCE. During RCE #1 subjects will also receive two biotinylated aliquots (~7 ml each) of RBCs drawn from the full INTERCEPT RBC unit before and after the PR process. The volume of each transfused aliquot will be assessed by weighing the syringe before and after transfusion. Each aliquot will be labeled at different biotin concentrations: (6 or 18 μg) to allow differentiation by flow cytometry. Subjects will be followed through a total of 4 sequential RCE episodes. Subjects will receive a full unit of INTERCEPT RBCs following RCE #2, with no biotinylated aliquots. No additional INTERCEPT RBCs will be transfused during RCE #3 or RCE #4.

To measure RBC recovery and blood volume, subject blood samples will be collected at the following time points:

* RCEs #1 and #2

  * Day 0: pre-RCE and at 15, 30, and 60 minutes post-RCE.
  * Days 1, 2-4, 7
  * Day 14 post-RCE #1 (no Day 14 sample after RCE #2).
* RCEs #3 and #4

  o Day 0: Fifteen minutes to 1 hour before and after the completion of each RCE episode.
* Appx Day 180 (±15 days) End of Study

Subjects will be screened for treatment-emergent antibodies to INTERCEPT RBCs and to biotinylated RBCs at screening and on day 14 post-RCE #1, Day 7 post-RCE #2, prior to RCE #3 and RCE #4 and on Day 180 (±15 days) post-RCE #1.

Subject RBC samples will be frozen and batched for flow-cytometry analysis at Cerus Corporation. De-glycerolized previously frozen RBCs will be used flow cytometry assessments. The assay to detect biotin levels by flow cytometry will use avidin- Allophycocyanin (APC) labeling in combination with an anti-acridine antibody. Acridine levels on INTERCEPT RBCs will be detected by flow cytometry utilizing a monoclonal antibody specific to the acridine moiety found on INTERCEPT RBCs. The antibody signal will be resolved in the phycoerythrin (PE) channel. QuantiBRITE PE beads (QB-PE) will be used to generate quasi-quantitative data for acridine RBC surface antigen labelling.

Subjects will be monitored closely during the blood transfusion procedure by staff trained to detect adverse events with transfusion. Laboratory monitoring for events of special interest will occur for 4 weeks (for hemolytic transfusion reactions) after RCE#1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* homozygous sickle cell disease (HbSS) or Hemoglobin S-β-thalassemia (HbSβ0) SCD
* Receiving RCE for ≥3 months prior to enrollment and scheduled to undergo at least 4 sequential RCE episodes during the period of enrollment in the study

Exclusion Criteria:

* Anticipated cessation of RBC transfusion therapy in the next ≤2 months
* Planned stem cell transplant or gene therapy in the next 6 months
* Delayed hemolytic transfusion reaction in the past 3 months
* History of hyperhemolysis syndrome at any time
* Consuming high-dose biotin or raw egg supplements
* Current pregnancy
* Antibody specific to INTERCEPT RBCs or biotinylated red blood cells (BioRBCs) at baseline
* Patients with RBC alloantibodies that make it difficult to provide antigen matched blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Recovery | 24 hour
  The volume of distribution and 24-hour post transfusion recovery (PTR24) of the INTERCEPT RBC units
Correlation between the biotin and acridine markers | 6 months
  Correlation between the biotin and acridine markers for determining the number of circulating INTERCEPT RBCs
Survival | 6 months
  Comparison of Pre-PR and INTERCEPT RBC PTR24, and survival over the duration of the study with intervening RCE procedures
Acridine loss | 6 months
  Kinetics of acridine loss from the INTERCEPT RBC surface

SECONDARY OUTCOMES:
Adverse Events | 6 months
  All subjects will be monitored for adverse events and transfusion reactions according to standard operating procedures at the RCE site
Treatment emergent antibodies | 6 months
  Safety assessments will also include screening for treatment emergent antibodies with specificity for INTERCEPT RBCs and for biotinylated RBCs on day 14 post-RCEs #1, Day 7 post-RCE #2, prior to RCE #3 and RCE #4 and on Day 180 (±15 days) post-RCE #1